CLINICAL TRIAL: NCT05624684
Title: Diagnostic Performance and Impact of a Multiplex PCR Pneumonia Panel on the Early Adaptation of Antimicrobial Therapy in ICU Patients With Severe Pneumonia. A Prospective Multicentric Observational Study.
Brief Title: Diagnostic Performance and Impact of a Multiplex PCR Pneumonia Panel in ICU Patients With Severe Pneumonia.
Status: Completed | Type: Observational
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Younes Aissaoui, MD, Professor of Anesthesiology and Intensive Care Medicine - Head of surgical intensive care unit, Avicenna Military Hospital
Other Study IDs: MORICUP-PCR study
Record Dates: First submitted 2022-11-04; First posted 2022-11-22 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Community-acquired Pneumonia; Hospital-acquired Pneumonia; Ventilator Associated Pneumonia
Keywords: Community-acquired Pneumonia; Hospital-acquired Pneumonia; Ventilator Associated Pneumonia; Multiplex PCR; Antibiotic stewardship
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ICU patients with severe pneumonia: Critically ill patients with severe pneumonia under mechanical ventilation including ventilator-associated pneumonia, community-acquired or hospital-acquired pneumonia.
  Interventions: Diagnostic Test: Multiplex respiratory PCR

INTERVENTIONS:
Diagnostic Test: Multiplex respiratory PCR — The BIOFIRE® FILMARRAY® Pneumonia plus Panel

SUMMARY:
The objective of this study is to assess the diagnostic performance of multiplex respiratory PCR (PCR-RM) compared to standard microbiological tests and its potential impact on the early adaptation of antibiotic treatment in intensive care patients with severe pneumonia.

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter ICU study. Adult patients with severe pneumonia requiring invasive mechanical ventilation will be included. Severe pneumonia consists of 3 categories of pneumonia: community-acquired pneumonia (CAP), hospital-acquired pneumonia (HAP), and ventilator-acquired pneumonia (VAP). The microbiological testing will be performed before antibiotic initiation on tracheobronchial aspirations, protected distal sampling, or mini-bronchoalveolar lavage as part of routine care. No additional samples will becollected for this study. Respiratory samples will be simultaneously tested by conventional microbiological techniques and multiplex respiratory PCR [PCR-RM] (BIOFIRE® FILMARRAY® Pneumonia Panel Plus). Classical microbiological culture (CMC) will be considered the gold standard for microbiological pneumonia diagnosis. The agreement between the results of the Pneumonia Plus® panel and the results of conventional microbial culture (CMC) will be assessed.

An empiric antibiotic therapy will be prescribed according to the local ecology and the protocols of each ICU unit. Two senior experts in each participating center will have to approve the antibiotic prescription. The antibiotic therapy could be modified after the reception of the Mutilpex PCR results by the two senior experts. After the reception of the results of the classic microbiological culture, the previous antibiotic changes will be judged as appropriate or inappropriate by a multidisciplinary team including intensivists, infectious disease specialists, and microbiologists. Appropriate changes include adequacy, de-escalation, and optimization of antibiotic therapy, and inappropriate changes include inadequacy, escalation, and de-optimization.

ELIGIBILITY:
Inclusion Criteria:

* critically ill adult patients
* clinical, biological, and radiological signs of severe pneumonia.
* community-acquired pneumonia, hospital-acquired pneumonia, or ventilator-associated pneumonia
* invasive mechanical ventilation.

Exclusion Criteria:

- Non-invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with ventilator-associated pneumonia (VAP), community-acquired pneumonia (CAP), or hospital-acquired pneumonia (HAP). For CAP and HAP, only patients under invasive mechanical ventilation will be included.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
The rate of diagnostic concordance between Classical microbiological cultures and the respiratory multiplex PCR (RM-PCR) and conventional microbiological cultures (CMC) to identify pathogens responsible for severe pneumonia in critically ill patients. | through study completion, an average of 6 months
  Classical microbiological cultures (CMC) will serve as the gold standard for the comparison between techniques, considering a test result:
  1. A true positive, when CMC and RM-PCR have identified the same microorganism (CMC+, PCR-RM +).
  2. A false positive, when RM-PCR detected an organism but not CMC (CMC-, RM-PCR+)
  3. A true negative, when no method detected any microorganism (CMC-, RM-PCR -)
  4. A false negative, when CMC but not RM-PCR has detected an organism (CMC+, RM-PCR -).
  Sensitivity, specificity, and positive and negative predictive values for the respiratory multiplex PCR will be calculated using the precedent findings.
The impact of the respiratory multiplex PCR (RM-PCR) on the appropriateness of empirical antimicrobial therapy. | through study completion, an average of 6 months
  The proportion of patients for whom the respiratory multiplex PCR (RM-PCR) induces an appropriate change of antibiotic therapy. Appropriate changes include adequacy, de-escalation, and escalation of antibiotic treatment.
  * Adequacy is defined as introducing an antibiotic to cover a microorganism that was not adequately treated before the results of RM-PCR.
  * Escalation is defined by a widening of the ATB spectrum to cover a pathogen not taken into account or the detection of resistance genes.
  * De-escalation is defined as the use of a narrower-spectrum anti-infective or the discontinuation of an ATB combination.

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenna Military Hospital, Marrakesh, Marrakesh Tensift El Haouz, Morocco

IPD SHARING:
Plan to Share IPD: Yes
The datasets of the study will be available from the principal investigator on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: until 5 years after study completion
Access Criteria: Healthcare workers.